CLINICAL TRIAL: NCT07335679
Title: Characterization of the Strasbourg Cohort of Patients With Adrenal Cortex Carcinoma
Acronym: CCSTR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9693
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Adrenal Cortical Carcinoma
Keywords: Adrenal cortical carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adrenal corticosteroid carcinoma (ACC) is a rare tumor of the adrenal cortex, with an estimated prevalence of 0.5 to 2 cases per million inhabitants per year.

Two peaks in incidence have been described: during the first decade of life and between 40 and 50 years of age, with a slight female predominance (female-to-male ratio of 1.5). The majority of cases (>90%) are sporadic, particularly in adults.

ACC may be discovered incidentally during an imaging examination performed for another reason (10 to 20% of cases) or in connection with a tumor syndrome (40-60% of cases) or hormonal hypersecretion (40 to 74% of cases). The diagnosis of CCS can be suggested by the combination of morphological characteristics seen on imaging and clinical and biological features (secretory syndrome), but only histopathology allows for a definitive diagnosis. Furthermore, histopathology enables the assessment of aggressiveness criteria (Weiss score, Ki67), which will influence further management and prognosis.

Given that CCS is a rare tumor, the investigators aim to study the clinical, biological, morphological, and histological characteristics and evaluate the prognosis of patients treated at our center in order to better understand the natural history of CCS and improve patient management.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥ 18 years old)
* Subjects followed at Strasbourg University Hospital for adrenal cortical carcinoma diagnosed between January 1, 2000, and May 31, 2025

Exclusion Criteria:

- Tumor reclassified as non-SCC by histopathology

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Adult subject (≥ 18 years old) followed at Strasbourg University Hospital for adrenal cortical carcinoma diagnosed between January 1, 2000, and May 31, 2025
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
Overall, specific, and progression-free survival in patients treated for adrenal cortical carcinoma (ACC) | Up to 12 months
  Overall survival:
  Is how long patients live after being diagnosed or treated, regardless of the cause of death.
  Example: If 100 patients are treated for ACC and 60 are alive after 5 years, the 5-year overall survival is 60%. It counts everyone, whether they die from ACC or something else, like an accident or another illness.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Endocrinologie, Diabétologie, Nutrition - CHU de Strasbourg - France, Strasbourg, France